CLINICAL TRIAL: NCT03857828
Title: Seminal Level of Clusterin in Infertile Men as a Predictor for Spermatogenesis Before Testicular Sperm Extraction
Brief Title: Seminal Level of Clusterin Before Testicular Sperm Extraction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Azza Sheshaey Hassan Abdelfadel Ahmad, Principal investigator, Assiut University
Other Study IDs: CLu before TESE
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Azoospermia, Nonobstructive
MeSH Terms: conditions — Azoospermia, Nonobstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: semen sample — • seminal sample for measuring clusterin level.

SUMMARY:
Measurement of clusterin level in the semen of infertile males undergoing testicular sperm extraction.

DETAILED DESCRIPTION:
Clusterin, known as apolipoprotein J, sulphated glycoprotein-2 or testosterone - repressed prostate message-2.

It plays important roles in several pathophysiological processes, including tissue remodelling, lipid transport, reproduction, complement regulation and apoptotic cell death .

As clusterin expression is markedly upregulated in various normal and malignant tissues undergoing apoptosis, it has been regarded as a marker for cell death.

There is a conflicting findings concerning the relationship between elevated clusterin expression and enhanced induction of apoptosis; that is, clusterin has appeared to have a powerful anti-apoptotic function through a chaperone-like activity.

In addition to the anti-apoptotic activity, seminal clusterin was reported to promote a tolerogenic response to male antigens, thereby contributing to female tolerance to seminal antigens.

In the testis, clusterin is secreted by Sertoli cells into the fluid of the seminiferous epithelium and deposited onto the membranes of elongating spermatids and mature spermatozoa.

To date, however, there has been little information with respect to the functional roles of clusterin in the male reproductive tract under physiological conditions.

In particular, it remains controversial as to whether or not clusterin helps assist the normal spermatogenesis.

Nonobstructive azoospermia (NOA) males are characterised by impaired spermatogenesis.

Although NOA patients have impaired global spermatogenic function, focal areas of spermatogenesis may still exist in their testes.

Focal spermatogenesis could possibly be obtained by testicular sperm extraction (TESE) technique .

A number of factors have been suggested to be of predictive value for patients with a good chance to retrieve sperm cell such as testicular volume, serum FSH levels , serum total testosterone and serum inhibin B levels.

ELIGIBILITY:
Inclusion Criteria:

* Infertile males , Azoospermia undergoing TESE as a preliminary step for ICSI .
* Age: 20-50 year

Exclusion Criteria:

* males <20 years and >50years
* Cryptorchidism .
* Testicular Agenesis and testicular atrophy .

Ages: 20 Years to 50 Years | Sex: Male
Age Groups: Adult
Gender Based: Yes
Study Population: Infertile Male patients (20 - 50 years ) with azoospermia undergoing testicular sperm extraction
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2020-12-16 (Estimated); Primary Completion 2020-12-16 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
The level of seminal clusterin before testicular sperm Extraction. | 1 hour
  Measurement of seminal clusterin by enzyme-linked immunosorbent assay (ELISA) and correlate them with the outcome of testicular sperm extraction to recognize predictors for spermatogenesis before testicular sperm extraction.